CLINICAL TRIAL: NCT00717470
Title: A Multicenter, Four Arm, Randomized, Open Label Clinical Study Investigating Optimized Dosing in a Prograf®-/Advagraf®-Based Immunosuppressive Regimen in Kidney Transplant Subjects (OSAKA Study)
Brief Title: A Study in Kidney Transplant Subjects to Investigate the Optimal Suppression of Immunity to Help Prevent Kidney Rejection
Acronym: OSAKA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PMR-EC-1210; 2007-005376-13 (EudraCT Number)
Record Dates: First submitted 2008-07-16; First posted 2008-07-17 (Estimated); Last update posted 2024-11-01 (Actual); Status verified 2024-10

CONDITIONS: Kidney Transplantation
Keywords: Kidney; Prograf; Transplant; Advagraf; Immunosuppression; FK506
MeSH Terms: interventions — Tacrolimus; Mycophenolic Acid; Basiliximab; Methylprednisolone; Prednisone; Adrenal Cortex Hormones

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Prograf + MMF + Steroids (Active Comparator): oral
  Interventions: Drug: Prograf®; Drug: Mycophenolate Mofetil; Drug: methylprednisolone / prednisone
- Advagraf (dose 1) + MMF + steroids (Active Comparator): oral
  Interventions: Drug: Advagraf®; Drug: Mycophenolate Mofetil; Drug: methylprednisolone / prednisone
- Advagraf (dose 2) + MMF + steroids (Active Comparator): oral
  Interventions: Drug: Advagraf®; Drug: Mycophenolate Mofetil; Drug: methylprednisolone / prednisone
- Advagraf + MMF + Basilixmab + steroids (Active Comparator): oral
  Interventions: Drug: Advagraf®; Drug: Mycophenolate Mofetil; Drug: Simulect; Drug: methylprednisolone / prednisone

INTERVENTIONS:
Drug: Prograf® — oral
  Other Names: FK506; Tacrolimus
  Arms: Prograf + MMF + Steroids
Drug: Advagraf® — oral
  Other Names: MR4; FK506XL; Tacrolimus extended release
  Arms: Advagraf (dose 1) + MMF + steroids; Advagraf (dose 2) + MMF + steroids; Advagraf + MMF + Basilixmab + steroids
Drug: Mycophenolate Mofetil — oral
  Other Names: MMF
Drug: Simulect — oral
  Other Names: basiliximab
  Arms: Advagraf + MMF + Basilixmab + steroids
Drug: methylprednisolone / prednisone — oral
  Other Names: corticosteroids

SUMMARY:
To compare how well the new formulation of Tacrolimus® used once daily, in combination with other drugs helps prevent the rejection of a new kidney after transplantation compared to the twice daily dose of Tacrolimus

ELIGIBILITY:
Inclusion Criteria:

* End stage kidney disease and a suitable candidate for primary renal transplantation or re-transplantation (unless the graft was lost from rejection within 12 months)
* Receiving a kidney transplant from a cadaveric or living (non HLA identical) donor with compatible ABO blood type
* Female subject of childbearing potential must have a negative serum pregnancy test at enrollment and must agree to maintain effective birth control during the study

Exclusion Criteria:

* Receiving or having previously received an organ transplant other than a kidney
* Cold ischemia time of the donor kidney > 30 hours
* Receiving a graft from a non-heart-beating donor other than of Maastricht category 3 (withdrawn of support awaiting cardiac arrest)
* Significant liver disease, defined as having continuously elevated SGPT/ALT and/or SGOT/AST and/or total bilirubin levels ≥ 2 times the upper value of the normal range of the investigational site or is receiving a graft from a hepatitis C or B positive donor
* Requiring initial sequential or parallel therapy with immunosuppressive antibody preparation(s)
* Requiring ongoing dosing with a systemic immunosuppressive drug prior to transplantation.
* Significant, uncontrolled concomitant infections and/or severe diarrhea, vomiting, active upper gastro-intestinal tract malabsorption or active peptic ulcer
* Pregnant woman or breast-feeding mother
* Subject or donor known to be HIV positive
* Known allergy or intolerance to tacrolimus, macrolide antibiotics, corticosteroids, basiliximab or mycophenolate mofetil or any of the product excipients
* Diagnosis of new-onset malignancy prior to transplantation, with the exception of basocellular or squamous cell carcinoma of the skin which had been treated successfully
* Currently participating in another clinical trial, and/or has taken an investigational drug within 28 days prior to enrollment
* Any form of substance abuse, psychiatric disorder or condition which, in the opinion of the investigator, may complicate communication with the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1252 (Actual)
Dates: Start 2008-05-14 (Actual); Primary Completion 2010-03-02 (Actual); Study Completion 2010-03-02 (Actual)

PRIMARY OUTCOMES:
Efficacy failure rate | 24 weeks

SECONDARY OUTCOMES:
Renal Function, acute rejection, Biopsy confirmed acute rejection | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Central Contact, Study Chair — Astellas Pharma Europe B.V.
Locations (102):
- Argentina (2):
  - Buenos Aires
  - Córdoba
- Austria (3):
  - Innsbruck
  - Linz
  - Vienna
- Belgium (3):
  - Brussels
  - Ghent
  - Leuven
- Czechia (4):
  - Brno
  - Hradec Kravlove
  - Ostrava
  - Prague
- France (18):
  - Angers
  - Bordeaux
  - Brest
  - Créteil
  - La Tronche
  - Le Kremlin-Bicêtre
  - Limoges
  - Lyon
  - Nantes
  - Nice
  - Paris
  - Rennes
  - Saint-Etienne
  - Strasbourg
  - Suresnes
  - Toulouse
  - Tours
  - Vandœuvre-lès-Nancy
- Germany (17):
  - Aachen
  - Berlin
  - Essen
  - Frankfurt
  - Freiburg I. Br
  - Halle
  - Hamburg
  - Hanover
  - Jena
  - Kaiserslautern
  - Kiel
  - Leipzig
  - München
  - Münster
  - Regensburg
  - Rostock
  - Tübingen
- Greece (2):
  - Athens
  - Thessaloniki
- Hungary (2):
  - Budapest
  - Szeged
- Dublin, Ireland
- Italy (7):
  - Ancona
  - Bologna
  - Milan
  - Padua
  - Roma
  - Siena
  - Treviso
- Maastricht, Netherlands
- Oslo, Norway
- Poland (6):
  - Bialystok
  - Gdansk
  - Lublin
  - Poznan
  - Warsaw
  - Wroclaw
- Portugal (2):
  - Lisbon
  - Porto
- Romania (2):
  - Bucharest
  - Cluj-Napoca
- Russia (4):
  - Moscow
  - Omsk
  - Saint Petersburg
  - Volgograd
- Slovakia (2):
  - Banska Bysterica
  - Košice
- South Africa (2):
  - Cape Town
  - Johannesburg
- Spain (16):
  - A Coruña
  - Albacete
  - Alicante
  - Barakaldo-Vizcaya
  - Barcelona
  - Cadiz
  - Granada
  - Madrid
  - Murcia
  - Oviedo
  - Palma de Mallorca
  - Pamplona
  - Salamanca
  - Seville
  - Valencia
  - Zaragoza
- Sweden (2):
  - Stockholm
  - Uppsala
- Zurich, Switzerland
- United Kingdom (4):
  - Birmingham
  - Glasgow
  - Leicester
  - Manchester

IPD SHARING:
Plan to Share IPD: Yes
Access to anonymized individual participant level data collected during the study, in addition to study-related supporting documentation, is planned for studies conducted with approved product indications and formulations, as well as products terminated during development. Studies conducted with product indications or formulations that remain active in development are assessed after study completion to determine if Individual Participant Data can be shared. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Access to participant level data is offered to researchers after publication of the primary manuscript (if applicable) and is available as long as Astellas has legal authority to provide the data.
Access Criteria: Researchers must submit a proposal to conduct a scientifically relevant analysis of the study data. The research proposal is reviewed by an Independent Research Panel. If the proposal is approved, access to the study data is provided in a secure data sharing environment after receipt of a signed Data Sharing Agreement.
URL: https://www.clinicaltrials.astellas.com/transparency/

REFERENCES:
- [Background] Albano L, Banas B, Klempnauer JL, Glyda M, Viklicky O, Kamar N; Optimising immunoSuppression After Kidney transplantation with ADVAGRAF Study Group. OSAKA trial: a randomized, controlled trial comparing tacrolimus QD and BD in kidney transplantation. Transplantation. 2013 Nov 27;96(10):897-903. doi: 10.1097/TP.0b013e3182a203bd. PMID 23982340
- [Derived] Kramer BK, Albano L, Banas B, Charpentier B, Backman L, Tedesco-Silva H Jr, Lehner F, Mondragon-Ramirez GA, Glyda M, Cassuto-Viguier E, Viklicky O, Mourad G, Rigotti P, Schleibner S, Kamar N. Efficacy of Prolonged- and Immediate-release Tacrolimus in Kidney Transplantation: A Pooled Analysis of Two Large, Randomized, Controlled Trials. Transplant Proc. 2017 Nov;49(9):2040-2049. doi: 10.1016/j.transproceed.2017.07.011. PMID 29149958
- See also: Link to results on Astellas Clinical Study Results website — https://www.astellasclinicalstudyresults.com/study.aspx?ID=58